CLINICAL TRIAL: NCT02437266
Title: Effect of Scapular Mobilization on Patients With Scapular Pain Associated With Myofascial Trigger Point
Brief Title: Effect of Scapular Mobilization on Patients With Scapular Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Vitsarut Buttagat, Dr. Vitsarut Buttagat, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55218152-5
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scapular mobilization (Experimental): The participants will receive a twenty minutes session of scapular mobilization onto the scapular
  Interventions: Other: Scapular mobilization
- Control (No Intervention): Rest on the bed for twenty minutes

INTERVENTIONS:
Other: Scapular mobilization
  Arms: Scapular mobilization

SUMMARY:
The purpose of this study is to determine the effect of scapular mobilization on pain related parameters including pain intensity, pressure pain threshold, muscle tension, anxiety, Scapular range of motion, patient satisfaction in patients with scapular pain associated with myofascial trigger point:

ELIGIBILITY:
Inclusion Criteria:

* The participants have experienced spontaneous scapular pain for longer than 12 weeks (chronic) and that at least one trigger point will be present in the muscles surrounding the scapula. Trigger points will be diagnosed as the presence of focal tenderness in a taut band and with pain recognition.
* The participants will be able to follow instructions.
* Good communication and cooperation.

Exclusion Criteria:

* Shoulder impingement syndrome
* Adhesive capsulitis
* Shoulder instability
* Shoulder arthritides
* Shoulder dislocation and/or bone fracture
* Hypermobility of shoulder joint
* Open wound
* Drug and/or alcohol intoxication
* Contraindications of mobilization

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Pain score on Visual analog scale | 5 weeks
  The intensity of pain will be reported by the participant on a visual analog scale ranging from 0 to 10. Zero indicates no pain anywhere and 10 indicates the most pain ever experienced.

SECONDARY OUTCOMES:
Pressure Pain Threshold as a measure by pressure algometry | 5 weeks
Anxiety on State Anxiety Inventory | 5 weeks
Scapular range of motion | 5 weeks
Patient satisfaction level | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Science, Mae Fah Luang University, Mueang, Changwat Chiang Rai, Thailand